CLINICAL TRIAL: NCT02205749
Title: Preferred Consent Models for Secondary Uses of Biospecimens Among Diverse Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 201208079; 3U54CA153460-03S1 (NIH)
Record Dates: First submitted 2014-07-29; First posted 2014-07-31 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Biospecimen Donation
Keywords: biobanks; informed consent; health literacy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Study-specific consent model (Other): • Review plain language brochure describing consent to a biobank based on the study-specific model of consent
  Interventions: Behavioral: Study-specific consent model; Behavioral: Broad consent model; Behavioral: Notice consent model
- Broad consent model (Other): • Review plain language brochure describing consent to a biobank based on the broad model of consent
  Interventions: Behavioral: Study-specific consent model; Behavioral: Broad consent model; Behavioral: Notice consent model
- Notice consent model (Other): • Review plain language brochure describing consent to a biobank based on the notice model of consent
  Interventions: Behavioral: Study-specific consent model; Behavioral: Broad consent model; Behavioral: Notice consent model

INTERVENTIONS:
Behavioral: Study-specific consent model — • Review plain language brochure describing consent to a biobank based on the study-specific model of consent
Behavioral: Broad consent model — • Review plain language brochure describing consent to a biobank based on the broad model of consent
Behavioral: Notice consent model — • Review plain language brochure describing consent to a biobank based on the notice model of consent

SUMMARY:
Research with stored biospecimens can provide substantial societal benefits, including greater understanding of cancer etiology and discovery of new cancer therapies, but one critical social and ethical issue is the use of samples for research unplanned at the time of biospecimen collection. Various models for consent (i.e., no consent, notice, opt-out, broad consent, study-specific consent) have been proposed for secondary research use of biospecimens, but empirical data on individuals' preferences for different consent models are limited, particularly from those with limited health literacy and from racial and ethnic minority groups. It is critically important to understand the consent preferences of diverse individuals, as participation of all population subgroups in biobanks is essential to reach translational cancer research goals. Based on a social ecological conceptual framework, the investigators will examine preferences for consent models for secondary research uses of biospecimens among a racially and socioeconomically diverse sample of women 35 years of age and older. The investigators aim to compare experimentally the effect of consent model on intentions to donate biospecimens for future research use among a diverse sample of women. The investigators hypothesize that women will have stronger intentions to donate based on the broad model of consent and the study-specific model of consent compared with the notice model of consent. These findings from groups underrepresented in research will be critical since the participation of these groups in biobanks is essential to generating findings that will achieve translational research goals of eliminating cancer disparities.

ELIGIBILITY:
Inclusion Criteria:

* 35 years old or older
* Proficient in English
* Identifies as Non-Hispanic
* Identifies as African-American or Black
* Identifies as Caucasian or White
* Identifies as Female

Exclusion Criteria:

* Under 35 years old
* Not proficient in English
* Identifies as Hispanic
* Identifies as a race other than African-American or Black; or Caucasian or White
* Identifies as more than one race
* Identifies as Male

Min Age: 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2013-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Intent to Donate | Immediate
  Intention to donate to a biobank.

SECONDARY OUTCOMES:
Consent Model Preference | Immediate
  Preferred type of consent for secondary use of biospecimens.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly A Kaphingst, ScD, Principal Investigator — The University of Utah; Bettina Drake, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine in St. Louis, St Louis, Missouri, United States